CLINICAL TRIAL: NCT06776380
Title: Pubertal Development in Patients with RASopathies
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: SN_PUBERTA2023
Record Dates: First submitted 2024-12-03; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-10

CONDITIONS: RASopathy
Keywords: RASopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Retrospective, single-centre, non-profit, observational study on pubertal development in patients with RASopathies.

Literature data shows that puberty can be delayed by about 2 years in patients with RASopathies and this has been associated with a reduced peak growth rate. To date, only a few numerically limited case series without molecular characterisation have been published.

This descriptive study should improve knowledge of pubertal development and its influence on growth and final stature. The primary aims are to describe the age of onset and progression of pubertal development in the cohort of patients with RASopathies, both male and female, and to describe the influence of pubertal development on statural growth and final stature in the same cohort.

DETAILED DESCRIPTION:
The study enrolls patients with molecularly confirmed RASopathy and completed pubertal development who referred to the Centre for Rare Congenital-Malformative Diseases of the Pediatrics Unit, IRCCS Azienda Ospedaliero-Universitaria di Bologna, Italy, between 01/01/2001 and 31/12/2023. Being a Regional Centre, it is possible to enrol a significant number of patients.

The primary aims of the study are to describe the age of onset and progression of pubertal development in this cohort of patients, and to describe the influence of pubertal development on statural growth and final stature. The secondary aim is to compare the trends of pubertal development and statural growth at puberty in GH-treated and untreated patients with RASopathies.

The study consists of the retrospective collection and analysis of anthropometric data on growth and pubertal development of the cohort of patients enrolled by consulting their medical records. More in detail, for each patient will be collected demographic data, prenatal data, personal medical history, pubertal history, organ involvement data, outpatient clinical evaluation with height, weight, and growth rate, data on GH therapy, if any, radiological assessments and laboratory tests, and the molecular RASopathy diagnosis by NGS panel and/or Sanger sequencing of target genes.

Due to the observational nature of the study, enrolled patients are treated according to clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Age at enrollment between 8 and 35 years, extremes included;
* Molecularly confirmed clinical diagnosis of RASopathy;
* Complete pubertal development;
* Obtaining informed consent for participation in the study and processing of personal data.

Exclusion Criteria:

• None.

Ages: 8 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients referred to the Pediatrics Unit of the IRCCS Azienda Ospedaliero-Universitaria di Bologna, Italy, between 01/01/2001 and 31/12/2023 with molecularly confirmed RASopathy and completed pubertal development.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-07-25 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Age of pubertal onset in males and females in all different genotypes | at baseline
  years, months
Proportion of males and females with delayed puberty in all different genotypes | at baseline
  percentage %
Age at the time of the presence of dosable serum LH (≥0,1 U/L) in males and females in all different genotypes | at baseline
  years, months
Age at time of presence of dosable serum estradiol (>15 pg/ml) in females in all different genotypes | at baseline
  years, months
Age at time of presence of dosable serum testosterone (>0,2 ng/ml) in males in all different genotypes | at baseline
  years, months
Age of reaching Peak Height Velocity in males and females in all different genotypes | at baseline
  years, months
Statural gain at puberty in males and females in all different genotypes | at baseline
  cm
Peak Height Velocity in males and females in all different genotypes | at baseline
  cm/year

SECONDARY OUTCOMES:
Height at first evaluation, final height, and statural gain at puberty in GH-treated and non-treated patients | at baseline
  cm
Peak Height Velocity in GH-treated and non-treated patients | at baseline
  cm/year
Age of reaching Peak Height Velocity in GH-treated and non-treated patients | at baseline
  years, months

CONTACTS AND LOCATIONS:
Overall Officials: Federica Tamburrino, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna, Italy